CLINICAL TRIAL: NCT05084222
Title: Use of Buventol Easyhaler and Bufomix Easyhaler as Relievers in Methacholine Challenge Testing and Inspiratory Flow Profiles During Induced Bronchoconstriction in Adult Subjects
Brief Title: Use of Buventol Easyhaler and Bufomix Easyhaler in Methacoline Challenge Testing
Acronym: EASYRELIEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0010032
Record Dates: First submitted 2021-09-15; First posted 2021-10-19 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buventol® Easyhaler® 200 µg/inhalation dmDPI (Experimental): 400 μg of salbutamol from Buventol Easyhaler is administered as two inhalations.
  Interventions: Drug: Buventol® Easyhaler® 200 µg/inhalation dmDPI
- Bufomix® Easyhaler® 160/4.5 µg/inhalation dmDPI (Experimental): 320 μg of budesonide and 9 μg of formoterol are administered from Bufomix Easyhaler as two inhalations.
  Interventions: Drug: Bufomix® Easyhaler® 160/4.5 µg/inhalation dmDPI
- Ventoline® Evohaler® 100 µg/inhalation pMDI (Active Comparator): 400 μg of salbutamol from Ventoline Evohaler is administered via Volumatic spacer as four inhalations.
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI

INTERVENTIONS:
Drug: Buventol® Easyhaler® 200 µg/inhalation dmDPI — Two doses will be administered
  Other Names: Salbutamol 200 µg/dose dmDPI
  Arms: Buventol® Easyhaler® 200 µg/inhalation dmDPI
Drug: Bufomix® Easyhaler® 160/4.5 µg/inhalation dmDPI — Two doses will be administered
  Other Names: Budesonide/formoterol 160/4.5 µg/inhalation dmDPI
  Arms: Bufomix® Easyhaler® 160/4.5 µg/inhalation dmDPI
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI — Four doses will be administered via Volumatic spacer
  Other Names: Salbutamol 100 µg/dose MDI
  Arms: Ventoline® Evohaler® 100 µg/inhalation pMDI

SUMMARY:
The study compares Buventol® Easyhaler® and Bufomix® Easyhaler® to the current standard treatment during methacholine challenge test. The trial will also provide inspiratory flow profile data for Easyhaler inhaler.

This trial is designed to provide a further evidence for the use of Easyhaler in diagnostic bronchial challenge tests and on the use of Easyhaler inhaler during obstructive event.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Finnish speaking adult (≥ 18 years old) subject indicated for methacholine challenge test.
3. The subject experiences FEV1 drop ≥ 20% compared to post-diluent spirometry.

Exclusion Criteria:

1. Subjects not eligible for methacholine challenge test for example for any of the following reasons:

   * Any respiratory infection within 2 weeks, or severe respiratory infection within 4 weeks before the study visit
   * FEV1 < 60% of predicted or < 1.0 l
   * Inability to perform acceptable and repeatable spirometry manoeuvres throughout the test procedure
   * Uncontrolled hypertension
   * Acute chest pain or unstable angina pectoris
   * Significant cardiac arrhythmias
   * Pneumothorax or recent bronchoscopy
   * Myocardial infarction or stroke in last 3 months
   * Known aortic aneurysm
   * Recent eye surgery or intracranial pressure elevation risk
   * Cholinesterase inhibitor medication
   * Pregnant or lactating females
2. Subjects who have used the following treatments before the study visit:

   * Short-acting β-agonists within 12 h
   * Long-acting β-agonists within 36 h
   * Ultra-long-acting β-agonists within 48 h
   * Long-acting anti-muscarinic agents within 168 h
   * Short-acting anticholinergics within 12 h
   * Oral theophylline within 24 h
   * Inhaled corticosteroids, leukotriene receptor antagonists and chromones within 4 weeks
3. Known hypersensitivity to the active substance(s) or the excipients of the study treatments (for example severe milk allergy, lactose contains small amounts of milk protein).
4. Administration of another investigational medicinal product within 30 days before the study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 10 minutes
  Mean change in FEV1 from post-diluent to FEV1 after the first dose of reliever.

SECONDARY OUTCOMES:
Number of subjects who recover from bronchoconstriction after first dose | 10 minutes
  Proportion of the subjects who recover to FEV1 > -10% compared to post-diluent FEV1 after first dose of reliever.
Forced expiratory volume in one second (FEV1) | 10 minutes
  Relative recovery of FEV1 after the study treatment dosing when compared to post-diluent FEV1.
Number of subjects who recover from bronchoconstriction after second dose | 20 minutes
  Proportions of subjects reaching FEV1 > -10% of post-diluent value after second dose of reliever.

OTHER OUTCOMES:
Number of patients needing medical attention | After study treatment administration until study completion (an average of 2.5 hours)
  Proportion of subjects needing medical attention after study treatment
Inhalation profile via Easyhaler | Before methacholine challenge and 10 minutes after the subject experiences FEV1 drop ≥ 20% compared to post-diluent spirometry
  Time-inspiratory flow -curve via Easyhaler measured with spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Lehtimäki, Principal Investigator — Tampere University Hospital, Finland
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No